CLINICAL TRIAL: NCT04290429
Title: Analysis of the Effect of Teduglutide Treatment on Intestinal Malabsorption and Paneth Cell Numbers in Patients With Steroid-refractory Gastrointestinal Graft Versus Host Disease (SR-GI-GVHD).
Brief Title: Treatment of Patients With Teduglutide (GLP-2) for GVHD and Analysis of Paneth Cells of GVHD Patients
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Freiburg (Other)
Responsible Party: Principal Investigator, Robert Zeiser, Director of the Division of Tumor Immunology, University of Freiburg
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GLP-2 in GVHD
Record Dates: First submitted 2020-02-26; First posted 2020-03-02 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Graft Versus Host Disease
MeSH Terms: conditions — Graft vs Host Disease | interventions — teduglutide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- SR-GI-GVHD (Experimental): Analysis of patient's stool frequency, albumin serum levels and quantification of Paneth cell numbers in GI biopsies before and during teduglutide treatment.
  Interventions: Drug: Teduglutide

INTERVENTIONS:
Drug: Teduglutide — Treatment of patients with SR-GI-GVHD with teduglutide

SUMMARY:
In this study the investigators evaluate the outcomes of six steroid-refractory GVHD patients with gastrointestinal signs of GVHD that were treated with teduglutide.

DETAILED DESCRIPTION:
Preliminary studies have showed that Glucagon-like peptide 2 (GLP-2) has regenerative and protective effects on the gastrointestinal tract after bowel injury. It induces positive effects in the GI tract like nutrient uptake, mucosal growth, protection from inflammation, etc. One of the target organs from GVHD is the GI tract, and since patients suffering from GI-GVHD experience intestinal disorders like loss of mucosal epithelial integrity, diarrhea accompanied by strong abdominal pain that can lead to food inanition, the investigators therefore aimed to examine the outcome of patients suffering from SR-GI-GVHD that are treated with the GLP-2 analogue, Teduglutide. The investigators will determine the outcome of each patient by monitoring the gastrointestinal signs like diarrhea frequency, intestinal absorption measured by serum-albumin concentrations and GI histology, specifically the number of Paneth cells before and during teduglutide treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with signs of acute SR-GI-GVHD
* Age ≥ 18 years
* Peripheral blood and stool samples available before and during treatment
* Written informed consent
* Ability to understand the nature of the study and the study related procedures and to comply with them

Exclusion Criteria:

* Age ≤ 18 years
* Lack of informed consent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2017-12-06 (Actual); Primary Completion 2019-12-06 (Actual); Study Completion 2019-12-06 (Actual)

PRIMARY OUTCOMES:
Paneth cell numbers | 2 years
  Quantification of Paneth cell numbers within the intestinal crypts before and during teduglutide treatment.

SECONDARY OUTCOMES:
Stool frequency | 2 years
  Analysis of patient's stool frequency before and during teduglutide treatment.
Intestinal absorption | 2 years
  Analysis of patient's albumin serum levels before and during teduglutide treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Zeiser, Prof. Dr., Principal Investigator — Medical Center University of Freiburg
Locations (1):
- Medical Center University of Freiburg, Freiburg im Breisgau, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zeiser R, Blazar BR. Acute Graft-versus-Host Disease - Biologic Process, Prevention, and Therapy. N Engl J Med. 2017 Nov 30;377(22):2167-2179. doi: 10.1056/NEJMra1609337. No abstract available. PMID 29171820
- [Background] Drucker DJ, Yusta B. Physiology and pharmacology of the enteroendocrine hormone glucagon-like peptide-2. Annu Rev Physiol. 2014;76:561-83. doi: 10.1146/annurev-physiol-021113-170317. Epub 2013 Oct 25. PMID 24161075
- [Background] Drucker DJ, Erlich P, Asa SL, Brubaker PL. Induction of intestinal epithelial proliferation by glucagon-like peptide 2. Proc Natl Acad Sci U S A. 1996 Jul 23;93(15):7911-6. doi: 10.1073/pnas.93.15.7911. PMID 8755576
- [Background] Boushey RP, Yusta B, Drucker DJ. Glucagon-like peptide (GLP)-2 reduces chemotherapy-associated mortality and enhances cell survival in cells expressing a transfected GLP-2 receptor. Cancer Res. 2001 Jan 15;61(2):687-93. PMID 11212269
- [Background] Jeppesen PB, Hartmann B, Thulesen J, Graff J, Lohmann J, Hansen BS, Tofteng F, Poulsen SS, Madsen JL, Holst JJ, Mortensen PB. Glucagon-like peptide 2 improves nutrient absorption and nutritional status in short-bowel patients with no colon. Gastroenterology. 2001 Mar;120(4):806-15. doi: 10.1053/gast.2001.22555. PMID 11231933
- [Background] Jeppesen PB, Pertkiewicz M, Messing B, Iyer K, Seidner DL, O'keefe SJ, Forbes A, Heinze H, Joelsson B. Teduglutide reduces need for parenteral support among patients with short bowel syndrome with intestinal failure. Gastroenterology. 2012 Dec;143(6):1473-1481.e3. doi: 10.1053/j.gastro.2012.09.007. Epub 2012 Sep 11. PMID 22982184